CLINICAL TRIAL: NCT00430638
Title: A Double-Blind, Randomized, Placebo Controlled, Parallel Group Study to Compare the Safety and Efficacy of an Olmesartan Medoxomil Based Treatment Regimen to Placebo in Patients With Stage I and Stage II Hypertension
Brief Title: A Study of the Blood Pressure Lowering Ability and Safety of Olmesartan Medoxomil in Stage I and Stage II Hypertension
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Daiichi Sankyo (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 866-451
Record Dates: First submitted 2007-02-01; First posted 2007-02-02 (Estimated); Results first posted 2010-01-22 (Estimated); Last update posted 2018-10-02 (Actual); Status verified 2018-09

CONDITIONS: Hypertension
Keywords: Hypertension; Angiotensin Receptor Blocker; Calcium Channel Blocker; Angiotensin Converting Enzyme Inhibitor; Hydrochlorothiazide; Stage I and II Hypertension
MeSH Terms: conditions — Hypertension | interventions — Olmesartan Medoxomil; Hydrochlorothiazide

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (2):
- Treatment (Experimental): Olmesartan medoxomil, plus hydrochlorothiazide, if necessary
  Interventions: Drug: olmesartan medoxomil + hydrochlorothiazide, if necessary
- Placebo (Placebo Comparator): Placebo tablets were taken once daily for 12 weeks
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: olmesartan medoxomil + hydrochlorothiazide, if necessary — olmesartan medoxomil + hydrochlorothiazide, if necessary. Oral tablets administered for once daily for 12 weeks
  Arms: Treatment
Drug: Placebo — Oral tablets administered for once daily for 12 weeks
  Arms: Placebo

SUMMARY:
This 16 week study will examine the ability of olmesartan medoxomil to lower the blood pressure of patients with moderate to severe high blood pressure in comparison to placebo. The medication being tested has been approved by the FDA for the treatment of high blood pressure.

DETAILED DESCRIPTION:
This study was to randomize an equal number of participants to either an olmesartan medoxomil based treatment or to placebo. The titration scheme was as follows:

* First 3 weeks (wks), all participants - olmesartan medoxomil 20 mg or placebo
* Next 3 wks, participants whose blood pressure was not controlled - olmesartan medoxomil 40 mg or placebo
* Next 3 wks, participants whose blood pressure was not controlled - olmesartan medoxomil 40 mg/HCT 12.5 mg or placebo
* Final 3 wks, participants whose blood pressure was not controlled - olmesartan medoxomil 40 mg/HCT 25 mg or placebo
* Subjects with a mean BP of <120/80 mmHg at any visit were considered responders and were not titrated up to the next dose level. However, they remained in the study at their currently assigned dose of study medication.
* Subjects with a mean office SBP ≥120 mmHg or a mean office DBP ≥80 mmHg at any subsequent visit(s) were considered 'uncontrolled' and were titrated to the next dose level according to the titration scheme above.
* Subjects who reach the highest dose (ie, olmesartan medoxomil 40 mg/HCT 25 mg) remained on that dose until study exit at Visit 8, unless safety concerns caused discontinuation of treatment.

ELIGIBILITY:
Inclusion Criteria:

* Greater than or equal to 18 years of age.
* Patients with a mean seated systolic blood pressure (MSSBP) greater than or equal to 140 mmHg but less than or equal to 179 mmHg and a mean seated diastolic blood pressure (MSDBP) less than or equal to 109 mmHg following a 3 to 4-week single-blind placebo run-in period.
* The difference in MSSBP between Visits 3 and 4 or between Visits 4 and 4X must be less than or equal to 10 mmHg.
* Patients with a mean daytime (8AM-4PM) systolic blood pressure (SBP) greater than or equal to 135 mmHg and less than or equal to 179 mmHg and a mean daytime diastolic blood pressure (DBP) less than or equal to 109 mmHg as measured by an ambulatory blood pressure monitoring device (ABPM) following placebo run-in period.
* If female, must have negative serum pregnancy test at screening and be either post-menopausal (greater than or equal to 1 year), had a hysterectomy or tubal ligation at least 6 months before consent or if of childbearing potential, must practice approved measures of birth control throughout study.

Exclusion Criteria:

* History of stroke or transient ischemic attack (TIA) within the last one year.
* History of myocardial infarction, coronary angioplasty, coronary artery bypass graft, or heart failure within the past 6 months.
* Patients with secondary hypertension of any etiology, such as renal disease, pheochromocytoma, or Cushing's syndrome.
* Type I diabetes. Patients with Type II diabetes on stable treatment, with fasting glucose <160 mg/dl may enroll.
* Patients with hemodynamically significant cardiac valvular disease.
* Patients with clinically significant cardiac conduction defects, including first, second or third degree AV block, left bundle branch block, sick sinus syndrome, atrial fibrillation, atrial flutter, an accessory bypass tract, or any arrhythmia requiring medication.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 278 (Actual)
Dates: Start 2006-12; Primary Completion 2007-10 (Actual); Study Completion 2007-10 (Actual)

CONTACTS AND LOCATIONS:
Locations (29):
- United States (29):
  - Birmingham, Alabama
  - Mobile, Alabama
  - Muscle Shoals, Alabama
  - Searcy, Arkansas
  - Carmichael, California
  - Spring Valley, California
  - Coral Gables, Florida
  - Deerfield Beach, Florida
  - DeLand, Florida
  - Fort Lauderdale, Florida
  - Hialeah, Florida
  - Hollywood, Florida
  - Pembroke Pines, Florida
  - Chicago, Illinois
  - Elizabeth, New Jersey
  - Winston-Salem, North Carolina
  - Cincinnati, Ohio
  - Oklahoma City, Oklahoma
  - Eugene, Oregon
  - Downingtown, Pennsylvania
  - Charleston, South Carolina
  - Nashville, Tennessee
  - New Tazewell, Tennessee
  - Colleyville, Texas
  - San Antonio, Texas
  - Murray, Utah
  - Manassas, Virginia
  - Olympia, Washington
  - Madison, Wisconsin

REFERENCES:
- [Result] Kereiakes DJ, Maa JF, Shojaee A, Dubiel R. Effect of an olmesartan medoxomil-based treatment algorithm on systolic blood pressure in patients with stage 1 or 2 hypertension: a randomized, double-blind, placebo-controlled study. Am J Cardiovasc Drugs. 2010;10(4):239-46. doi: 10.2165/11538630-000000000-00000. PMID 20653330
- [Result] Oparil S, Chrysant SG, Kereiakes D, Xu J, Chavanu KJ, Waverczak W, Dubiel R. Results of an olmesartan medoxomil-based treatment regimen in hypertensive patients. J Clin Hypertens (Greenwich). 2008 Dec;10(12):911-21. doi: 10.1111/j.1751-7176.2008.00045.x. PMID 19120717

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects were recruited at 29 US sites (private medical practices and small clinics) over 5 months from December 2006 to May 2007 from each physician's clientele base. About 450 potential subjects were to be screened so that about 250 eligible subjects, men and women at least 18 years of age with stage I or II hypertension, were randomized.
Pre-assignment Details: After 3-4 weeks of placebo treatment, eligible subjects were randomized. 140 were randomized to drug; 138 to placebo. 2 active drug participants were given the wrong dose at entry. Because only 138 participants received Olmesartan 20 mg, any demography data totals are equal to 276 instead of 278. The subgroup analyses are similarly affected.
Groups:
- Placebo (Pbo) Group: 138 were randomized to placebo. Participants remained in the placebo group for the duration of the study. The study medication was titrated at 3-week intervals if blood pressure goals were not achieved. The medications were: all started on placebo matching olmesartan 20 mg; after 3 weeks, if necessary, placebo matching olmesartan 40 mg; after 6 weeks, if necessary, placebo matching olmesartan 40 mg + hydrochlorothiazide 12.5 mg; after 9 weeks, if necessary, placebo matching olmesartan 40 mg + hydrochlorothiazide 25 mg.
- Olmesartan Group: 140 participants were randomized to the olmesartan group. These participants remained in this group for the entire study. The study medication was titrated at 3-week intervals if blood pressure goals were not achieved. The medications were: all started on olmesartan 20 mg; after 3 weeks, if necessary, olmesartan 40 mg; after 6 weeks, if necessary, olmesartan 40 mg + hydrochlorothiazide 12.5 mg; after 9 weeks, if necessary, olmesartan 40 mg + hydrochlorothiazide 25 mg.
Period: Overall Study
Arm/Group | Placebo (Pbo) Group | Olmesartan Group
Started | 138 | 140 (2 participants were erroneously assigned to olmesartan 40 mg instead of 20 mg)
Completed | 60 | 92
Not Completed | 78 | 48
Not completed — Adverse Event | 15 | 15
Not completed — Uncontrolled blood pressure | 48 | 13
Not completed — Lost to Follow-up | 1 | 7
Not completed — Protocol Violation | 6 | 4
Not completed — Withdrawal by Subject | 4 | 6
Not completed — Non-compliant | 2 | 1
Not completed — Other | 2 | 2

BASELINE CHARACTERISTICS:
Groups:
- Olmesartan Group: Participants were randomized to an olmesartan (Olm) based active treatment group. After 3,6,and 9 weeks of treatment participants were titrated to the next regiment if their blood pressure was greater than 120/80 mmHg. The active treatment group received olm 20 mg (weeks 1-3), olm 40 mg (weeks 4-6), olm 40 mg + 12.5 mg hydrchlorothiazide (HCTZ) (weeks 7-9), and olm 40 mg + 25 mg HCTZ (weeks 10-12).
- Placebo Group: Participants were randomized to a placebo (Pbo) group. The Pbo participants remained in the pbo group for the entire 12 weeks of treatment.
- Total: Total of all reporting groups
Arm/Group | Olmesartan Group | Placebo Group | Total
Number analyzed (Participants) | 138 | 138 | 276
Age, Continuous [Mean (Full Range); unit: years] | 55.9 (10.74) [26 to 86] | 55.8 (9.47) [35 to 80] | 55.9 (10.1) [26 to 86]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 75 | 72 | 147
  Male | 63 | 66 | 129
Region of Enrollment [Number; unit: participants]
  United States | 138 | 138 | 276
Diastolic BP [Mean (Full Range); unit: mm Hg] | 94.2 (7.7) [74 to 106] | 93.7 [69 to 107] | 94.0 [69 to 107]
Heart Rate [Mean (Full Range); unit: Beats/minute] | 75.1 (10.84) [52 to 122] | 73.6 [47 to 94] | 74.4 [47 to 122]
Systolic BP [Mean (Full Range); unit: mm Hg] | 156.9 (9.19) [140 to 178] | 155.4 [136 to 178] | 156.2 [136 to 178]

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Mean Systolic Blood Pressure (SBP) After 12 Weeks of Randomized Treatment as Measured by Omron Device.
Description: The change from baseline in mean systolic blood pressure (SBP) after 12 weeks of randomized treatment was compared between the olmesartan based treatment group and the placebo treatment group.
Time Frame: baseline to 12 weeks
Population: The efficacy cohort is defined as any subject who received at least 1 dose of randomized study medication and had a baseline and at least 1 post-baseline efficacy blood pressure assessment. 140 participants were originally randomized to the olmesartan group. 139 is the correct number analyzed. For the placebo group the efficacy cohort = 137.
Measure: Least Squares Mean (Standard Error); unit: mm Hg
Groups:
- Placebo: Patient received placebo tablets.
- Olmesartan Group: Participants received olmesatan medoxomil plus hydrochlorothiazide, if necessary.
Arm/Group | Placebo | Olmesartan Group
Number analyzed (Participants) | 137 | 139
mm Hg | -0.1 (1.40) | -22.3 (1.39)
Statistical Analysis 1: Comparison: Placebo vs Olmesartan Group; Null hypothesis: For the entire efficacy population, Olmesartan had the same effect on change from baseline in systolic blood pressure at week 12 as Placebo. A statistical test was evaluated at the 2 sided significance level of 5% without adjustment for multiple comparisons; Test type: Superiority or Other; p < 0.0001, ANCOVA — No multiplicity adjustments; The ANCOVA model included randomized treatment and baseline cuff blood pressure stage as factors and study baseline systolic BP value as a covariate

2. Secondary Outcome: Change From Baseline in Mean Diastolic Blood Pressure (DBP) After 12 Weeks of Randomized Treatment as Measured by Omron Device.
Description: Change from study baseline (average of triplicate DBP measurements at the last 2 qualifying visits during placebo run-in period) in DBP to the end of 12 weeks of randomized treatment using a last observation carried forward (LOCF) approach.
Time Frame: baseline to 12 weeks
Population: The efficacy cohort is defined as any subject who received at least 1 dose of randomized study medication and had a baseline and at least 1 post-baseline efficacy blood pressure assessment. 140 participants were originally randomized to the olmesartan group, but two were erroneously started with the 40mg dose. 139 is the correct number analyzed.
Measure: Least Squares Mean (Standard Error); unit: mm Hg
Groups:
- Placebo Group: Patient received placebo tablets throughout the 12-week active treatment period.
- Olmesartan Group: Participants received olmesartan medoxomil tablets + hydrochlorothiazide tablets, if necessary, once daily for the duration of the 12-week active treatment period.
Arm/Group | Placebo Group | Olmesartan Group
Number analyzed (Participants) | 137 | 139
mm Hg | -0.8 (0.78) | -12.1 (0.77)
Statistical Analysis 1: Comparison: Placebo Group vs Olmesartan Group; Null hypothesis: For the entire efficacy population, Olmesartan had the same effect on change from baseline in diastolic blood pressure at week 12 as Placebo. A statistical test was evaluated at the 2 sided significance level of 5% without adjustment for multiple comparisons; Test type: Superiority or Other; p < 0.0001, ANCOVA; The ANCOVA Model included randomized treatment and baseline cuff BP stage as factors and study baseline diastolic BP as a covariate

3. Secondary Outcome: The Difference in the Change From Baseline to Week 12 in Seated Systolic and Diastolic Blood Pressure Between the Olmesartan Group and the Placebo Group for Males.
Description: The difference in the change from baseline to week 12 in seated systolic and diastolic blood pressure for males in the olmesartan group vs. the placebo group was analyzed.
Time Frame: Baseline to week 12
Population: 131 male participants
Measure: Least Squares Mean (Standard Error); unit: mm Hg
Arm/Group | Olmesartan vs. Placebo
Number analyzed (Participants) | 131
mm Hg
  Systolic Blood Pressure | -22.6 (2.94)
  Diastolic Blood Pressure | -13.5 (1.66)
Statistical Analysis 1: Comparison: Olmesartan vs. Placebo; Null hypothesis (male systolic blood pressure (SBP)): For the male efficacy population, Olmesartan had the same effect on change from baseline in systolic blood pressure at week 12 as Placebo. A statistical test was evaluated at the 2 sided significance level of 5% without adjustment for multiple comparisons; Test type: Superiority or Other; p < 0.0001, ANCOVA
Statistical Analysis 2: Comparison: Olmesartan vs. Placebo; Null hypothesis (Males - diastolic blood pressure (DBP)): For the male efficacy population, Olmesartan had the same effect on change from baseline in diastolic blood pressure at week 12 as Placebo. A statistical test was evaluated at the 2 sided significance level of 5% without adjustment for multiple comparisons; Test type: Superiority or Other; p < 0.0001, ANCOVA

4. Secondary Outcome: The Difference in the Change From Baseline to Week 12 in Seated Systolic and Diastolic Blood Pressure Between the Olmesartan Group and the Placebo Group for Females.
Description: The difference in the change from baseline to week 12 in seated blood pressure for females in the olmesartan group vs. the placebo group was analyzed.
Time Frame: Baseline to week 12
Population: 145 female participants from both the olmesartan and placebo groups were analyzed.
Measure: Least Squares Mean (Standard Deviation); unit: mm Hg
Groups:
- Olmesartan vs. Placebo: 145 females participants were analyzed.
Arm/Group | Olmesartan vs. Placebo
Number analyzed (Participants) | 145
mm Hg
  Systolic blood pressure | -21.6 (2.6)
  Diastolic blood pressure | -12.0 (1.38)
Statistical Analysis 1: Comparison: Olmesartan vs. Placebo; Null hypothesis (Systolic blood pressure (SBP) - females): For the female efficacy population, Olmesartan had the same effect on change from baseline in systolic blood pressure at week 12 as Placebo. A statistical test was evaluated at the 2 sided significance level of 5% without adjustment for multiple comparisons; Test type: Superiority or Other; p < 0.0001, ANCOVA
Statistical Analysis 2: Comparison: Olmesartan vs. Placebo; Null hypothesis (Diastolic blood pressure (DBP) - females): For the female efficacy population, Olmesartan had the same effect on change from baseline in DBP at week 12 as Placebo. A statistical test was evaluated at the 2 sided significance level of 5% without adjustment for multiple comparisons; Test type: Superiority or Other; p < 0.0001, ANCOVA

5. Secondary Outcome: The Difference in the Change From Baseline to Week 12 in Seated Systolic and Diastolic Blood Pressure Between the Olmesartan Group and the Placebo Group for Participants Less Than 65 Years Old.
Time Frame: Baseline to 12 weeks
Population: 232 participants from both the olmesartan and placebo groups, less than 65 years of age, were analyzed.
Measure: Least Squares Mean (Standard Deviation); unit: mm Hg
Arm/Group | Olmesartan vs. Placebo
Number analyzed (Participants) | 232
mm Hg
  Systolic blood pressure | -23.8 (2.04)
  Diastolic blood pressure | -13.6 (1.17)
Statistical Analysis 1: Comparison: Olmesartan vs. Placebo; Null hypothesis(Systolic blood pressure (SBP) - less than 65 years of age): For the efficacy population < 65 years of age, Olmesartan had the same effect on change from baseline in SBP at week 12 as Placebo. A statistical test was evaluated at the 2 sided significance level of 5% without adjustment for multiple comparisons; Test type: Superiority or Other; p < 0.0001, ANCOVA
Statistical Analysis 2: Comparison: Olmesartan vs. Placebo; Null hypothesis (Diastolic blood pressure (DBP) - less than 65 years of age): For the efficacy population < 65 years of age, Olmesartan had the same effect on change from baseline in DBP at week 12 as Placebo. A statistical test was evaluated at the 2 sided significance level of 5% without adjustment for multiple comparisons; Test type: Superiority or Other; p < 0.0001, ANCOVA

6. Secondary Outcome: The Difference in the Change From Baseline to Week 12 in Seated Systolic and Diastolic Blood Pressure Between the Olmesartan Group and the Placebo Group for Participants Greater Than or Equal to 65 Years Old.
Time Frame: Baseline to 12 weeks
Population: 44 participants of greater than 65 years of age, from both the olmesartan and placebo groups were analyzed.
Measure: Least Squares Mean (Standard Deviation); unit: mm Hg
Arm/Group | Olmesartan vs. Placebo
Number analyzed (Participants) | 44
mm Hg
  Systolic blood pressure | -16.1 (6.18)
  Diastolic blood pressure | -9.0 (2.42)
Statistical Analysis 1: Comparison: Olmesartan vs. Placebo; Null hypothesis (Systolic blood pressure (SBP) - > or equal to 65 years old): For the efficacy population > or = to 65 years of age, Olmesartan had the same effect on change from baseline in SBP at week 12 as Placebo. A statistical test was evaluated at the 2 sided significance level of 5% without adjustment for multiple comparisons; Test type: Superiority or Other; p = 0.0125, ANCOVA
Statistical Analysis 2: Comparison: Olmesartan vs. Placebo; Null hypothesis (Diastolic blood pressure (DBP) > or equal to 65): For the efficacy population > or = to 65 years of age, Olmesartan had the same effect on change from baseline in DBP at week 12 as Placebo. A statistical test was evaluated at the 2 sided significance level of 5% without adjustment for multiple comparisons; Test type: Superiority or Other; p = 0.0006, ANCOVA

7. Secondary Outcome: The Difference in the Change From Baseline to Week 12 in Seated Systolic and Diastolic Blood Pressure Between the Olmesartan Group and the Placebo Group for Black Participants.
Time Frame: Baseline to week 12
Population: 55 Black participants from both the olmesartan and placebo groups were analyzed.
Measure: Least Squares Mean (Standard Deviation); unit: mm Hg
Arm/Group | Olmesartan vs. Placebo
Number analyzed (Participants) | 55
mm Hg
  Systolic blood pressure | -21.3 (4.97)
  Diastolic blood pressure | -12.5 (2.72)
Statistical Analysis 1: Comparison: Olmesartan vs. Placebo; Null hypothesis (Systolic blood pressure (SBP) - Black participants): For the Black efficacy population, Olmesartan had the same effect on change from baseline in SBP at week 12 as Placebo. A statistical test was evaluated at the 2 sided significance level of 5% without adjustment for multiple comparisons; Test type: Superiority or Other; p < 0.0001, ANCOVA
Statistical Analysis 2: Comparison: Olmesartan vs. Placebo; Null hypothesis (Diastolic blood pressure (DBP) - Black participants): For the Black efficacy population, Olmesartan had the same effect on change from baseline in DBP at week 12 as Placebo. A statistical test was evaluated at the 2 sided significance level of 5% without adjustment for multiple comparisons; Test type: Superiority or Other; p < 0.0001, ANCOVA

8. Secondary Outcome: The Difference in the Change From Baseline to Week 12 in Seated Systolic and Diastolic Blood Pressure Between the Olmesartan Group and the Placebo Group for Non-Black Participants.
Time Frame: Baseline to 12 weeks
Population: 221 non-Black participants from both the olmesartan and placebo groups were analyzed.
Measure: Least Squares Mean (Standard Deviation); unit: mm Hg
Arm/Group | Olmesartan vs. Placebo
Number analyzed (Participants) | 221
mm Hg
  Systolic blood pressure | -22.3 (2.14)
  Diastolic blood pressure | -12.8 (1.18)
Statistical Analysis 1: Comparison: Olmesartan vs. Placebo; Null hypothesis(Systolic blood pressure (SBP) - non-Black participants): For the Non-Black efficacy population, Olmesartan had the same effect on change from baseline in SBP at week 12 as Placebo. A statistical test was evaluated at the 2 sided significance level of 5% without adjustment for multiple comparisons; Test type: Superiority or Other; p < 0.0001, ANCOVA
Statistical Analysis 2: Comparison: Olmesartan vs. Placebo; Null hypothesis(Diastolic blood pressure (DBP) - non-Black participants): For the Non-Black efficacy population, Olmesartan had the same effect on change from baseline in DBP at week 12 as Placebo. A statistical test was evaluated at the 2 sided significance level of 5% without adjustment for multiple comparisons; Test type: Superiority or Other; p < 0.0001, ANCOVA

9. Secondary Outcome: The Difference in the Change From Baseline to Week 12 in Seated Systolic and Diastolic Blood Pressure Between the Olmesartan Group and the Placebo Group for Stage 1 Hypertensives
Time Frame: Baseline to 12 weeks
Population: 130 Stage 1 hypertensive participants from both the olmesartan and placebo groups.
Measure: Least Squares Mean (Standard Deviation); unit: mm Hg
Arm/Group | Olmesartan vs. Placebo
Number analyzed (Participants) | 130
mm Hg
  Systolic blood pressure | -22.1 (2.43)
  Diastolic blood pressure | -12.2 (1.39)
Statistical Analysis 1: Comparison: Olmesartan vs. Placebo; Null hypothesis(Systolic blood pressure (SBP) - Stage 1 hypertensive participants): For the Stage 1 efficacy population, Olmesartan had the same effect on change from baseline in SBP at week 12 as Placebo. A statistical test was evaluated at the 2 sided significance level of 5% without adjustment for multiple comparisons; Test type: Superiority or Other; p < 0.0001, ANCOVA
Statistical Analysis 2: Comparison: Olmesartan vs. Placebo; Null hypothesis (Diastolic blood pressure (DBP) - Stage 1 hypertensive participants): For the Stage 1 efficacy population, Olmesartan had the same effect on change from baseline in DBP at week 12 as Placebo. A statistical test was evaluated at the 2 sided significance level of 5% without adjustment for multiple comparisons; Test type: Superiority or Other; p < 0.0001, ANCOVA

10. Secondary Outcome: The Difference in the Change From Baseline to Week 12 in Seated Systolic and Diastolic Blood Pressure Between the Olmesartan Group and the Placebo Group for Stage 2 Hypertensives
Time Frame: Baseline to 12 months
Population: 146 Stage 2 hypertensive participants from both the olmesartan and placebo groups
Measure: Least Squares Mean (Standard Deviation); unit: mm Hg
Arm/Group | Olmesartan vs. Placebo
Number analyzed (Participants) | 146
mm Hg
  Systolic blood pressure | -22.5 (3.07)
  Diastolic blood pressure | -13.2 (1.65)
Statistical Analysis 1: Comparison: Olmesartan vs. Placebo; Null hypothesis (Systolic blood pressure (SBP) - Stage 2 hypertensive participants): For the Stage 2 efficacy population, Olmesartan had the same effect on change from baseline in SBP at week 12 as Placebo. A statistical test was evaluated at the 2 sided significance level of 5% without adjustment for multiple comparisons; Test type: Superiority or Other; p < 0.0001, ANCOVA
Statistical Analysis 2: Comparison: Olmesartan vs. Placebo; Null hypothesis (Diastolic blood pressure (DBP) - Stage 2 hypertensive participants): For the Stage 2 efficacy population, Olmesartan had the same effect on change from baseline in DBP at week 12 as Placebo. A statistical test was evaluated at the 2 sided significance level of 5% without adjustment for multiple comparisons; Test type: Superiority or Other; p < 0.0001, ANCOVA

ADVERSE EVENTS:
Time Frame: 12-week randomized, treatment period plus 30 days after the last dose of study medication.
Description: All adverse events (whether observed by the Investigator or reported by the subject) were recorded on the Adverse Event page of the CRF with details of the following: date, time of onset, duration, severity, relationship to study drug, action taken with respect to the study drug, treatments administered, outcome, and seriousness.
Arm/Group | Placebo (Pbo) Group | Olmesartan Group
Serious Adverse Events (participants affected / at risk) | 0/138 | 3/140
Other Adverse Events (participants affected / at risk) | 46/138 | 55/140
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (Pbo) Group (N=138) | Olmesartan Group (N=140)
Hypertension (Vascular disorders) | 0 | 1
Small Intestine Obstruction (Gastrointestinal disorders) | 0 | 1
Supraventricular tachycardia (Cardiac disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (Pbo) Group (N=138) | Olmesartan Group (N=140)
Back pain (Musculoskeletal and connective tissue disorders) | 4 | 8
Cough (Respiratory, thoracic and mediastinal disorders) | 7 | 3
Dizziness (Nervous system disorders) | 1 | 13
Headache (Nervous system disorders) | 17 | 11
Hypertension (Vascular disorders) | 1 | 3
Seasonal allergy (Immune system disorders) | 2 | 3
Upper respiratory tract infection (Infections and infestations) | 7 | 9
Urinary tract infection (Infections and infestations) | 0 | 4
Viral upper respiratory infection (Infections and infestations) | 7 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
If identified by Daiichi Sankyo Inc.(DSI), any of DSI's confidential information, as defined to the author, shall be deleted. Nothing in our site agreement shall be taken as giving DSI any right of editorial control over any publication prepared by the study site.